CLINICAL TRIAL: NCT02858453
Title: The LEADERSHIP 301 Trial: A 12-Week, Randomized, Multi-Center, Double-Blind, Placebo-Controlled, 3-Arm, Parallel-Group, Phase 3 Trial to Evaluate the Efficacy and Safety of 2 Doses of AQX-1125 Targeting the Src Homology 2-containing Inositol-5'-Phosphatase 1 (SHIP1) Pathway in Subjects With Interstitial Cystitis/Bladder Pain Syndrome Followed by an Extension Period
Brief Title: Efficacy and Safety of 2 Doses of AQX-1125 in Subjects With Interstitial Cystitis / Bladder Pain Syndrome
Acronym: LEADERSHIP 301
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aquinox Pharmaceuticals (Canada) Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AQX-1125-301
Record Dates: First submitted 2016-04-19; First posted 2016-08-08 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Interstitial Cystitis; Bladder Pain Syndrome; Painful Bladder Syndrome; Chronic Interstitial Cystitis
Keywords: Interstitial cystitis; Bladder pain syndrome; Painful bladder syndrome; Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS); AQX-1125; SHIP1; Chronic interstitial cystitis
MeSH Terms: conditions — Cystitis, Interstitial | interventions — 4-(4-(aminomethyl)-7a-methyl-1-methylideneoctahydro-1H-inden-5-yl)-3-(hydroxymethyl)-4-methylcyclohexan-1-ol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AQX-1125 100 mg (Experimental): 2 tablets, by mouth, once per day for 12 weeks; followed by a 52-week Extension Period
  Interventions: Drug: AQX-1125 100 mg
- AQX-1125 200 mg (Experimental): 2 tablets, by mouth, once per day for 12 weeks; followed by a 52-week Extension Period
  Interventions: Drug: AQX-1125 200 mg
- Placebo (Placebo Comparator): 2 placebo tablets, by mouth, once per day for 12 weeks; followed by randomization to 100 mg or 200 mg AQX-1125 for a 52-week Extension Period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AQX-1125 100 mg — Synthetic SHIP1 activator
  Arms: AQX-1125 100 mg
Drug: AQX-1125 200 mg — Synthetic SHIP1 activator
  Arms: AQX-1125 200 mg
Drug: Placebo — Appearance and weight matched placebo tablets
  Arms: Placebo

SUMMARY:
This study evaluates the effects of two doses of oral AQX-1125 on bladder pain and other urinary symptoms in subjects with interstitial cystitis/bladder pain syndrome. Participants will receive either 100 mg AQX-1125, 200 mg AQX-1125 or placebo for the first 12 weeks of the study. After 12 weeks, all participants will receive either 100 mg or 200 mg AQX-1125 for 52 weeks.

DETAILED DESCRIPTION:
This multi-center Phase 3 trial includes a randomized, double-blind, placebo-controlled, parallel-group, treatment phase to evaluate the efficacy and safety of 2 doses of oral AQX-1125 in up to 600 subjects with interstitial cystitis/bladder pain syndrome.

The primary objective of this study is to evaluate the effect of 12 weeks of treatment of AQX-1125 (100 mg or 200 mg) administered once daily compared to placebo on the change from Baseline to Week 12 in maximum daily bladder pain using a standardized 11-point numerical rating scale pain score recorded daily by electronic diary (e-diary).

The 12-week Treatment Period is followed by an Extension Period of 52 weeks. Randomization and start of dosing occurs at Baseline and is followed by visits at Week 6 and Week 12. At the end of Week 12, subjects will be randomized into the 52-week Extension Period. Subjects on active treatment during the Treatment Period will continue on that same dose for the Extension Period, while subjects receiving placebo during the Treatment Period will be randomized to one of the active doses of 100 mg or 200 mg AQX-1125 for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female, ≥18 and ≤80 years of age who have had symptoms of bladder pain in addition to urinary urgency and/or urinary frequency for more than 6 months
* Have had a clinical diagnosis, or history consistent with the diagnosis, of interstitial cystitis/bladder pain syndrome for >3 months but ≤20 years
* Must be capable of voiding independently
* Have undergone a cystoscopy within the last 36 months prior to Baseline
* Women of child bearing potential must have a negative pregnancy test, be non-lactating and agree to avoid pregnancy and use a highly effective method of contraception with one additional barrier method of contraception from screening until at least 28 days after the last dose of study drug has been taken
* Men must use a condom for sexual intercourse from screening until at least 90 days after last dose of study drug has been taken, unless they have been surgically sterilized (vasectomy)

Exclusion Criteria

* Have had a urinary tract infection (UTI) including bacterial cystitis within the past 30 days
* Microscopic hematuria that has not been adequately evaluated as per local standard of care
* Have a history of chronic substance abuse, dependency or abuse of opiates, or other narcotics within the last 2 years
* History of previous procedure(s) (augmentation cystoplasty, cystectomy, cytolysis, botulinum toxin or bladder catheterization) that has significantly affected bladder function
* History of cyclophosphamide or chemical cystitis, urinary tuberculosis or radiation cystitis
* Women: History of bladder tumors; uterine, cervical, vaginal or urethral cancer
* Men: History of prostate surgery (transurethral resection of the prostate [TURP], transurethral resection tumor [TURT], transurethral incision of the prostate [TUIP], transurethral needle ablation [TUNA] etc.), a history of prostate cancer or currently being treated for chronic bacterial prostatitis
* Major surgery within 3 months prior to Screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Maximum Daily Bladder Pain Score | Baseline to 12 weeks
  Change from Baseline for AQX-1125 100 mg or 200 mg compared to placebo in the maximum daily bladder pain score based on a standardized 11-point numeric rating scale (NRS) recorded by electronic diary (e-diary)

SECONDARY OUTCOMES:
Change from Baseline in Voiding Frequency Measured Over a 24 hr Period | Baseline to 12 weeks
  Change from Baseline for AQX-1125 100 mg or 200 mg compared to placebo in voiding frequency measured over a 24-hour period
Change from Baseline Interstitial Cystitis Symptom Index Score | Baseline to 12 weeks
  Change from Baseline for AQX-1125 100 mg or 200 mg compared to placebo in Interstitial Cystitis Symptom Index Score
Change from Baseline in Bladder Pain/Interstitial Cystitis Symptom Score | Baseline to 12 weeks
  Change from Baseline for AQX-1125 100 mg or 200 mg compared to placebo in Bladder Pain/Interstitial Cystitis Symptom Score
Change from Baseline in Subject's Global Response Assessment | Baseline to 12 weeks
  Change from Baseline for AQX-1125 100 mg or 200 mg compared to placebo in subject's Global Response Assessment

OTHER OUTCOMES:
Frequency and Severity of Adverse Events | Baseline to 12-weeks; during 52-week EP and baseline to 64-weeks, with a 4-week post-dose, and 6 month post-dose (ocular only), follow-up
  Adverse events and abnormal clinically significant vital signs, laboratory tests, electrocardiogram, weight, physical examination findings and ophthalmological examination findings

CONTACTS AND LOCATIONS:
Overall Officials: Robert Moldwin, MD, Principal Investigator — Hofstra Northwell School of Medicine
Locations (119):
- United States (56):
  - Site 9035, Homewood, Alabama
  - Site 9026, Tucson, Arizona
  - Site 9064, Little Rock, Arkansas
  - Site 9010, Beverly Hills, California
  - Site 9060, Escondido, California
  - Site 9011, Los Angeles, California
  - Site 9021, Los Angeles, California
  - Site 9019, Los Angeles, California
  - Site 9023, Murrieta, California
  - Site 9015, Orange, California
  - Site 9039, Palo Alto, California
  - Site 9003, San Diego, California
  - Site 9046, Sherman Oaks, California
  - Site 9070, Whittier, California
  - Site 9004, Farmington, Connecticut
  - Site 9029, Middlebury, Connecticut
  - Site 9013, Noblesville, Indiana
  - Site 9049, West Des Moines, Iowa
  - Site 9054, Metairie, Louisiana
  - Site 9007, Shreveport, Louisiana
  - Site 9038, Owings Mills, Maryland
  - Site 9005, Boston, Massachusetts
  - Site 9028, Watertown, Massachusetts
  - Site 9034, Grand Rapids, Michigan
  - Site 9020, Royal Oak, Michigan
  - Site 9042, Troy, Michigan
  - Site 9072, Omaha, Nebraska
  - Site 9062, Cranford, New Jersey
  - Site 9001, Edison, New Jersey
  - Site 9025, Albuquerque, New Mexico
  - Site 9016, Brooklyn, New York
  - Site 9066, Cheektowaga, New York
  - Site 9037, New Hyde Park, New York
  - Site 9041, The Bronx, New York
  - Site 9068, Morehead City, North Carolina
  - Site 9002, Raleigh, North Carolina
  - Site 9055, Wilmington, North Carolina
  - Site 9045, Winston-Salem, North Carolina
  - Site 9058, Winston-Salem, North Carolina
  - Site 9048, Cleveland, Ohio
  - Site 9033, Cleveland, Ohio
  - Site 9047, Gahanna, Ohio
  - Site 9051, Toledo, Ohio
  - Site 9053, Oklahoma City, Oklahoma
  - Site 9071, Oklahoma City, Oklahoma
  - Site 9050, Bala-Cynwyd, Pennsylvania
  - Site 9031, Bryn Mawr, Pennsylvania
  - Site 9036, Newtown, Pennsylvania
  - Site 9032, Philadelphia, Pennsylvania
  - Site 9040, Greer, South Carolina
  - Site 9027, Franklin, Tennessee
  - Site 9069, Houston, Texas
  - Site 9030, Houston, Texas
  - Site 9052, Temple, Texas
  - Site 9012, Richmond, Virginia
  - Site 9008, Mountlake Terrace, Washington
- Belgium (3):
  - Site 1103, Edegem
  - Site 1102, Ghent
  - Site 1101, Roeselare
- Canada (10):
  - Site 1013, Kelowna, British Columbia
  - Site 1005, Brampton, Ontario
  - Site 1006, Burlington, Ontario
  - Site 1002, Kingston, Ontario
  - Site 1003, Kitchener, Ontario
  - Site 1015, Oakville, Ontario
  - Site 1010, Toronto, Ontario
  - Site 1017, Québec, Quebec
  - Site 1016, Sherbrooke, Quebec
  - Site 1008, Sherbrooke, Quebec
- Czechia (7):
  - Site 2002, Hradec Králové
  - Site 2006, Jablonec nad Nisou
  - Site 2003, Kolín
  - Site 2001, Pilsen
  - Site 2007, Prague
  - Site 2004, Prague
  - Site 2005, Uherské Hradiště
- Site 3002, Herlev, Denmark
- Hungary (3):
  - Site 4004, Budapest
  - Site 4001, Csongrád
  - Site 4003, Sopron
- Latvia (5):
  - Site 5005, Daugavpils
  - Site 5001, Jelgava
  - Site 5002, Liepāja
  - Site 5003, Riga
  - Site 5004, Riga
- Netherlands (2):
  - Site 1301, Rotterdam, South Holland
  - Site 1302, The Hague
- Poland (9):
  - Site 6011, Bydgoszcz
  - Site 6009, Gdynia
  - Site 6004, Gdynia
  - Site 6005, Piaseczno
  - Site 6001, Poznan
  - Site 6007, Poznan
  - Site 6002, Siedlce
  - Site 6008, Warsaw
  - Site 6003, Warsaw
- Romania (11):
  - Site 7007, Brasov
  - Site 7010, Bucharest
  - Site 7008, Bucharest
  - Site 7002, Bucharest
  - Site 7005, Bucharest
  - Site 7009, Bucharest
  - Site 7004, Bucharest
  - Site 7006, Craiova
  - Site 7011, Craiova
  - Site 7003, Sibiu
  - Site 7001, Târgu Mureş
- Spain (4):
  - Site 1401, Aravaca
  - Site 1402, Córdoba
  - Site 1405, Elche
  - Site 1403, Vic
- United Kingdom (8):
  - Site 8008, Plymouth, Devon
  - Site 8001, Sheffield, South Yorkshire
  - 8005, Coventry, Warwickshire
  - Site 8007, Wolverhampton, West Midlands
  - Site 8009, London
  - Site 8004, London
  - Site 8002, Reading
  - Site 8003, Wakefield